CLINICAL TRIAL: NCT02204670
Title: Exercise and Irisin Trial (EXIT): Prospective Cohort Study of the Determinants of the Metabolic Response to Exercise in Obese Adolescents
Brief Title: EXIT: Prospective Study of the Response to Exercise
Acronym: EXIT
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jon McGavock, Associate Professor Department of Pediatrics and Child Health, University of Manitoba
Other Study IDs: B2014:064
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Liver Fat; Type 2 Diabetes
Keywords: Irisin; Obesity; Exercise; Myokine; Impaired Glucose Tolerance
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus, Type 2; Obesity; Motor Activity; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Overweight Adolescents Performing Resistance Training: Overweight adolescents that meet pre-specified enrollment criteria will all undergo supervised resistance exercise for a 6-week period. Prior to training, all participants will undergo a single bout of resistance training to determine the acute release of Irisin with resistance training. This will be the primary exposure variable. After the acute session, all participants will perform resistance training three times per week for a period of 4 weeks. During each session participants will perform 3 sets of 8-12 repetitions (60-85% of 1RM) for major muscle groups (quadriceps, shoulders, and pectoral).
  Interventions: Other: Acute release of irisin after a single exercise session.

INTERVENTIONS:
Other: Acute release of irisin after a single exercise session. — We will determine the amount of Irisin secreted after a single bout of resistance exercise. Participants will be stratified into 3 groups based on the degree of Irisin release during this acute bout of resistance exercise. The metabolic adaptations to the 4 weeks of resistance training will be compared between youth stratified according to the amount of Irisin released during the acute bout of resistance exercise.

SUMMARY:
Background :

Regular exercise is a cornerstone in the prevention and the management of comorbidities. Unfortunately, the metabolic benefit of exercise training is not universal and varies among individuals. A main factor likely to explain the exercise training variability is the lack of empirical evidence on the determinants of exercise training. A series of muscle-derived cytokines have recently been discovered that (1) are released during exercise and (2) exert positive effects on peripheral tissues. Irisin is one of these novel "myokines" and might contributes to the metabolic adaptations to exercise training.

Methods:

The investigators will perform a pilot cohort study in which obese adolescents will perform resistance exercise training for 6 weeks. The main exposure variable will be the acute release of irisin during resistance exercise. The main outcome measures will be the change in hepatic triglyceride content and glucose area under the curve during a 75g, 2-hour oral glucose tolerance test.

Study Hypothesis:

The primary overall hypothesis is that the change in plasma Irisin with a single bout of exercise will be associated with the metabolic adaptations to 6 weeks of resistance training, specifically, the reductions in hepatic triglyceride content and post-prandial glucose excursions, in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents (12-18 years)
2. Body mass index considered obese according to the International Obesity Task Force

Exclusion Criteria:

1. Adolescents with medication-induced or type 1 diabetes
2. are currently being treated with corticosteroids or atypical antipsychotics, as these agents significantly influence carbohydrate metabolism
3. have an orthopaedic injury or chronic illness that would prevent them from performing the intervention
4. have experienced >10% weight loss or enrolled in weight loss program within six months of enrolment
5. a history of alcoholism or drug abuse
6. require use of medication(s) known to affect insulin sensitivity or secretion within the last 30 days
7. medication(s) known to cause weight gain
8. anabolic steroids
9. weight loss medication(s)
10. pregnant or planning to be pregnant

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A community-based convenient sample of overweight adolescents aged 12-18 years with a BMI > 95th centile for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Hepatic Triglyceride Content | 6 weeks
  Hepatic triglyceride content will be measured by using 1H magnetic resonance spectroscopy. After image acquisition, a single voxel volume of interest will be placed in the upper right lobe of the liver in an area devoid of adipose tissue to acquire 1H spectra. A total of 64 spectra will be collected and averaged to determine the intracellular triglyceride content.

SECONDARY OUTCOMES:
Post-prandial glucose | 6 weeks
  Glucose area under the curve (AUC) will be determined by summing the area under serum glucose measures between each 15- or 30-min segment using the trapezium rule during a frequently sampled 75-g oral glucose challenge .

CONTACTS AND LOCATIONS:
Overall Officials: Jon M McGavock, PhD, Principal Investigator — University of Manitoba
Locations (1):
- The Manitoba Institute of Child Health, Winnipeg, Canada